CLINICAL TRIAL: NCT06160141
Title: Effect of Two Years of Resistance Training in Cardiac Function in Older Women: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Edilson Serpeloni Cyrino, PhD, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GEPEMENE 2023
Record Dates: First submitted 2023-11-09; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Aging; Healthy
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Training groups vs. Control Group
Who Masked: Outcomes Assessor
Masking Description: Assessor was blind to the primary outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): The training group performed 48 weeks of resistance training, 3 times per week.
  Interventions: Other: Resistance training
- Control Group (No Intervention): The control group did not performed any kind of resistance exercises.

INTERVENTIONS:
Other: Resistance training — Resistance training program. The RT program was performed over 48 weeks, three times per week (Mondays, Wednesdays, and Fridays), during the morning, in the University fitness facility. Participants were personally supervised by Physical Education professionals (1-2 supervisors per exercise) with substantial RT experience to ensure consistent and safe exercise performance.
  Participants performed four exercises for the trunk and upper limbs and four exercises for the lower limbs in three sets of 8-12 repetitions. T Rest intervals were 1-2 and 2-3 min between sets and exercises. The training load was individually adjusted for each exercise weekly, according to the number of repetitions performed during the last training session, to ensure that the subjects kept performing at the ideal intensity for the repetition zone. In these situations, training loads were increased by 2-5% for upper-limb exercises and 5-10% for lower-limb exercises.
  Arms: Training group

SUMMARY:
Purpose: This study aimed to determine the effect of 48 weeks of resistance training (RT) on cardiac function in older women. Methods: Sixty-four older women (≥ 60 years), physically independent, were selected for this study. Participants were randomized into a training group (TG, n = 33) and a control group (CG, n = 31). The RT program was conducted over 48 weeks, three sessions a week, on nonconsecutive days, in the morning hours. Participants performed eight exercises for the whole body (chest press, horizontal leg press, seated row, leg extension, triceps pushdown, lying leg curl, preacher curl, seated calf raise) in three sets of 8-12 repetitions. The echocardiography was performed according to current guidelines before and after 48 weeks by an experienced echocardiographer blinded to patient status and group assignment. One-repetition maximum (1-RM) tests were used to analyze muscular strength. Glusoce, lipid profile, and C-reactive protein were measured. DEXA was used to measure body fat and muscle mass.

DETAILED DESCRIPTION:
Echocardiography exams were performed according to current guidelines, at baseline and the end of the study, by an experienced echocardiographer blinded to patient status and group assignment in a Philips ultrasound machine, model iE33 (Philips Medical Solutions, Noord Brabant, The Netherlands), equipped with S5-1 and X5-1 transducer. According to current recommendations, cardiac chamber dimensions, volumes, and left ventricular mass were measured. Mitral inflow velocities were assessed using pulsed-wave Doppler in the apical four-chamber view, with the sample volume placed between the tips of the mitral leaflets; velocities were recorded at end-expiration. Tissue Doppler velocities were acquired at end-expiration, in the apical four-chamber view, with the sample positioned at the septal and lateral mitral annulus for determination of systolic (S'), early diastolic (E'), and late diastolic (A') velocities. Pulsed wave Doppler velocities at the upper right pulmonary vein were also recorded. For all parameters, the average of three consecutive heartbeats was recorded.

Dietary intake - The 24-hour dietary recall method was used to analyze the participants' habitual intake throughout the study. Assessments were performed on three non-consecutive days of the week, in the first and last two weeks of each intervention phase. During the interviews, a photographic manual of food portion size was presented to the participants to improve the quality of food intake reports. Homemade measurements of the nutritional values of food were converted into grams and milliliters by the online software Virtual Nutri Plus (Keeple®, Rio de Janeiro, RJ, Brazil) for diet analysis. All foods not found in the program database were added to food tables.

Muscular strength Maximal dynamic strength was evaluated using one-repetition maximum (1RM) tests on the chest press, leg extension, and preacher curl exercises (Ipiranga Fitness, Presidente Prudente, SP, Brazil), respectively, following standard procedures 17,18. Three 1RM testing sessions were performed in the morning, separated by 48 h intervals. In each session, participants completed a warm-up of 10-15 repetitions before each exercise with approximately 50% of the estimated load to the first attempt, followed by three maximal attempts. For the first day of testing, the first selected load was based on the researchers' experience and perception of the difficulty (effort) with which participants performed the warm-up. If the first attempt was completed, the load was added for the subsequent attempts (3-10% of the previous effort). If an attempt was unsuccessful, load was removed in the same proportion. The rest period was three to five minutes between attempts and five minutes between exercises. The load for the first attempt in the second and third sessions was the maximal obtained in the previous session. Participants were encouraged to perform two repetitions with the selected load during each effort in the three exercises. The 1RM was recorded as the heaviest load lifted in which participants could complete only one voluntary muscle action among the three sessions. In addition, a total muscular strength score was calculated as the sum of the highest scores in each of the three exercises. Two experienced researchers supervised each exercise during testing sessions to standardize technique reliability and ensure the safety of participants.

Body composition. Dual-energy X-ray absorptiometry exams were performed in a Lunar Prodigy device, model NRL 41990 (General Electric, Madison, USA), to determine the total, regional lean soft tissue (LST), appendicular LST (ALST), and the total body, trunk, gynoid, and android fat masses. Participants were instructed to remove all metal objects before scanning to minimize possible estimation errors. Scans were performed with participants lying in the supine position along the table's longitudinal centerline axis. Feet were secured together at the toes to immobilize the legs while the hands were maintained in a pronated position within the scanning region. A skilled researcher carried out both calibration and analysis, following the manufacturer's recommendations. The software generated standard lines that separated the limbs from the trunk and head. The same technician adjusted these lines using specific anatomical points determined by the manufacturer and performed all analyses during the intervention. A predictive equation estimated total-body skeletal muscle mass from ALST.

Functional fitness tests - Four motor tests determined functional fitness: gait speed (4-m usual walking speed), walking agility, 30-s chair stand, and 6-min walk (6MWT). Three evaluators used stopwatches (KIKOS, São Paulo, SP, Brazil) to measure participants' time walking a 4-m usual walking speed. Adhesive tapes on the floor demarcated this distance with additional 2-m patches before and after the 4-m main patch. Participants walked 8-m, but only the time spent walking the middle 4-m was timed to the nearest 0.01 s. Participants completed three attempts, with the mean used for analysis. For the walking agility test, participants were seated on a chair supported by a wall, with their back in contact with the backrest, feet fully supported on the floor, and hands rested on the thighs. Participants were requested to stand up, walk around a cone at a distance of 2.44 m in front of the chair, return to the chair and sit down. Participants were instructed to complete the path as quickly as possible without running. Time was recorded to the nearest 0.01 s with a stopwatch from the initial movement to rise from the chair until returning to sit down again. Participants completed three trials, with the best one recorded for analysis. For the 30-s chair stand test, participants were seated on a chair supported by a wall, with their back in contact with the backrest, feet fully supported on the floor, and hands crossed to rest on their opposite shoulders. Participants performed the maximum sit-to-stand repetitions possible within 30 seconds. An evaluator recorded the time and counted the number of completed repetitions performed. For the 6MWT, each participant was instructed to walk as far as possible, without running, around a rectangular path (4.6 x 18.4 m, total perimeter: 46.0 m) marked with ribbons and cones on the floor for 6-min. An evaluator timed the test time, counted the number of laps, and calculated the total distance covered with an accuracy of one meter. The 6MWT assesses walking ability and endurance.

Metabolic biomarkers - The blood sample (venous) was collected in a tube containing a dipotassium ethylenediaminetetraacetic acid (12 ml, vacuum-sealed system; Vacutainer, England) between 7:00 and 9:00 a.m. by a trained laboratory technician after an overnight fast of at least 12 h. Participants rested in a seated position for at least five minutes before withdrawing 5 ml of blood from a prominent superficial vein in the antecubital space. All samples were centrifuged at 3,000 rpm for 15 min, and plasma or serum aliquots were stored at -80° C until assayed. As determined in human plasma, inter- and intra-assay coefficients of variation were < 10%. Measurements of serum levels of high-sensitivity C-reactive protein, glucose, total cholesterol (TC), high-density lipoprotein cholesterol (HDL-c), and triglycerides (TG) were determined by standard methods in a specialized laboratory at University Hospital. The low-density lipoprotein cholesterol (LDL-c) was calculated using the following equation: LDL-c = TC - (HDL-c + TG/5). The analyses were performed using a Dimension RxL Max biochemical auto-analyzer system (Siemens Dade Behring, Erlangen, Germany) according to established methods in the literature consistent with the manufacturer's protocol.

Resistance training program - The RT program was performed over 48 weeks, three times per week (Mondays, Wednesdays, and Fridays), during the morning, in the University fitness facility. Participants were personally supervised by Physical Education professionals (1-2 supervisors per exercise) with substantial RT experience to ensure consistent and safe exercise performance. Throughout the intervention period, the RT program was carried out on machines and free weights (Ipiranga Fitness, Presidente Prudente, SP, Brasil).

Participants performed four exercises for the trunk and upper limbs (chest press, seated row, triceps pushdown, preacher curl) and four exercises for the lower limbs (horizontal leg press, leg extension, lying leg curl, seated calf raise) in three sets of 8-12 repetitions. The participants were instructed to inhale during the eccentric phase and exhale during the concentric phase while maintaining a constant movement velocity at a ratio of approximately 1:2 s (concentric and eccentric muscle actions, respectively). Rest intervals were 1-2 and 2-3 min between sets and exercises. The training load was individually adjusted for each exercise weekly, according to the number of repetitions performed during the last training session, to ensure that the subjects kept performing at the ideal intensity for the repetition zone. In these situations, training loads were increased by 2-5% for upper-limb exercises and 5-10% for lower-limb exercises.

ELIGIBILITY:
Inclusion Criteria:

* females aged ≥ 60 years; physically independent; had no cardiac, orthopedic, or musculoskeletal dysfunction that could impede physical exercise; not having uncontrolled diabetes mellitus or hypertension; and not be involved in the practice of regular physical activity performed more than once a week over the three months before the start of the study

Exclusion Criteria:

* Not completed at least 80% of the sessions.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Doppler-echocardiography | 48 weeks
  Echocardiography exams were performed according to current guidelines, at baseline and the end of the study, by an experienced echocardiographer blinded to patient status and group. According to current recommendations, cardiac chamber dimensions, volumes, and left ventricular mass were measured. Mitral inflow velocities were assessed using pulsed-wave Doppler in the apical four-chamber view, with the sample volume placed between the tips of the mitral leaflets; velocities were recorded at end-expiration. Tissue Doppler velocities were acquired at end-expiration, in the apical four-chamber view, with the sample positioned at the septal and lateral mitral annulus for determination of systolic (S'), early diastolic (E'), and late diastolic (A') velocities. Pulsed wave Doppler velocities at the upper right pulmonary vein were also recorded. For all parameters, the average of three consecutive heartbeats was recorded.

SECONDARY OUTCOMES:
Dietary intake | 48 weeks
  The 24-hour dietary recall method was used to analyze the participants' habitual intake throughout the study. Assessments were performed on three non-consecutive days of the week, in the first and last two weeks of each intervention phase. During the interviews, a photographic manual of food portion size was presented to the participants to improve the quality of food intake reports. Homemade measurements of the nutritional values of food were converted into grams and milliliters by the online software Virtual Nutri Plus (Keeple®, Rio de Janeiro, RJ, Brazil) for diet analysis. All foods not found in the program database were added to food tables.
Muscular strength | 48 weeks
  Maximal dynamic strength was evaluated using one-repetition maximum (1RM) tests on the chest press, leg extension, and preacher curl exercises, respectively, following standard procedures. Three 1RM testing sessions were performed in the morning, separated by 48 h intervals. In each session, participants completed a warm-up of 10-15 repetitions before each exercise with approximately 50% of the estimated load to the first attempt, followed by three maximal attempts. For the first day of testing, the first selected load was based on the researchers' experience and perception of the difficulty (effort) with which participants performed the warm-up. If the first attempt was completed, the load was added for the subsequent attempts (3-10% of the previous effort).
Body composition | 48 weeks
  Dual-energy X-ray absorptiometry exams were performed in a Lunar Prodigy device, model NRL 41990 (General Electric, Madison, USA), to determine the total, regional lean soft tissue (LST), appendicular LST (ALST), and the total body, trunk, gynoid, and android fat masses. Participants were instructed to remove all metal objects before scanning to minimize possible estimation errors. Scans were performed with participants lying in the supine position along the table's longitudinal centerline axis. Feet were secured together at the toes to immobilize the legs while the hands were maintained in a pronated position within the scanning region. A skilled researcher carried out both calibration and analysis, following the manufacturer's recommendations.
Gait speed test | 48 weeks
  Three evaluators used stopwatches to measure participants' time walking a 4-m usual walking speed. Adhesive tapes on the floor demarcated this distance with additional 2-m patches before and after the 4-m main patch. Participants walked 8-m, but only the time spent walking the middle 4-m was timed to the nearest 0.01 s. Participants completed three attempts, with the mean used for analysis.
walking agility test | 48 weeks
  Participants were seated on a chair supported by a wall, with their back in contact with the backrest, feet fully supported on the floor, and hands rested on the thighs. Participants were requested to stand up, walk around a cone at a distance of 2.44 m in front of the chair, return to the chair and sit down. Participants were instructed to complete the path as quickly as possible without running. Time was recorded to the nearest 0.01 s with a stopwatch from the initial movement to rise from the chair until returning to sit down again. Participants completed three trials, with the best one recorded for analysis.
30-s chair stand test | 48 weeks
  Participants were seated on a chair supported by a wall, with their back in contact with the backrest, feet fully supported on the floor, and hands crossed to rest on their opposite shoulders. Participants performed the maximum sit-to-stand repetitions possible within 30 seconds. An evaluator recorded the time and counted the number of completed repetitions performed.
6-min walk (6MWT) | 48 weeks
  Each participant was instructed to walk as far as possible, without running, around a rectangular path (4.6 x 18.4 m, total perimeter: 46.0 m) marked with ribbons and cones on the floor for 6-min. An evaluator timed the test time, counted the number of laps, and calculated the total distance covered with an accuracy of one meter. The 6MWT assesses walking ability and endurance.
Serum levels of high-sensitivity C-reactive protein | 48 weeks
  The blood sample (venous) was collected in a tube containing a dipotassium ethylenediaminetetraacetic acid (12 ml, vacuum-sealed system; Vacutainer, England) between 7:00 and 9:00 a.m. by a trained laboratory technician after an overnight fast of at least 12 h. Participants rested in a seated position for at least five minutes before withdrawing 5 ml of blood from a prominent superficial vein in the antecubital space. The analyses were performed using a Dimension RxL Max biochemical auto-analyzer system.
Glucose | 48 weeks
  The blood sample (venous) was collected in a tube containing a dipotassium ethylenediaminetetraacetic acid (12 ml, vacuum-sealed system; Vacutainer, England) between 7:00 and 9:00 a.m. by a trained laboratory technician after an overnight fast of at least 12 h. Participants rested in a seated position for at least five minutes before withdrawing 5 ml of blood from a prominent superficial vein in the antecubital space. The analyses were performed using a Dimension RxL Max biochemical auto-analyzer system.
total cholesterol | 48 weeks
  The blood sample (venous) was collected in a tube containing a dipotassium ethylenediaminetetraacetic acid (12 ml, vacuum-sealed system; Vacutainer, England) between 7:00 and 9:00 a.m. by a trained laboratory technician after an overnight fast of at least 12 h. Participants rested in a seated position for at least five minutes before withdrawing 5 ml of blood from a prominent superficial vein in the antecubital space. The analyses were performed using a Dimension RxL Max biochemical auto-analyzer system.
high-density lipoprotein cholesterol (HDL-c) | 48 weeks
  The blood sample (venous) was collected in a tube containing a dipotassium ethylenediaminetetraacetic acid (12 ml, vacuum-sealed system; Vacutainer, England) between 7:00 and 9:00 a.m. by a trained laboratory technician after an overnight fast of at least 12 h. Participants rested in a seated position for at least five minutes before withdrawing 5 ml of blood from a prominent superficial vein in the antecubital space. The analyses were performed using a Dimension RxL Max biochemical auto-analyzer system.
triglycerides | 48 weeks
  The blood sample (venous) was collected in a tube containing a dipotassium ethylenediaminetetraacetic acid (12 ml, vacuum-sealed system; Vacutainer, England) between 7:00 and 9:00 a.m. by a trained laboratory technician after an overnight fast of at least 12 h. Participants rested in a seated position for at least five minutes before withdrawing 5 ml of blood from a prominent superficial vein in the antecubital space. The analyses were performed using a Dimension RxL Max biochemical auto-analyzer system.
low-density lipoprotein cholesterol (LDL-c) | 48 weeks
  The LDL-c was calculated using the following equation: LDL-c = TC - (HDL-c + TG/5).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual de Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No